CLINICAL TRIAL: NCT05951543
Title: Effects of Plyometric Exercises on Static and Dynamic Balance in Children With Down,s Syndrome
Brief Title: Effects of Plyometric Exercises on Static and Dynamic Balance of Children With Down,s Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0709
Record Dates: First submitted 2023-06-06; First posted 2023-07-19 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Down Syndrome
Keywords: Balance, Dynamic, Down syndrome, Plyometric, Static.
MeSH Terms: conditions — Down Syndrome | interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: It is a randomize control trail ,used to evaluate the effects of plyometric exercises on static and dynamic balance of children with down syndrome.subjects with down syndrome meeting the predetermine inclusion and exclusion criteria will be devided into two groups using simple random sampling technique.
Who Masked: Participant
Masking Description: participants will get separate treatment protocols and possible efferts will be put to mask the both groups about their treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plyometric group (Experimental): Experimental group will be given baseline exercises along with plyometric exercises such as Vertical jump, run and jump, drop jump (jump height between 40 and 50 cm) drop jump and horizontal jump with same height from 3rd week.particepents perform exercises carrying medicine balls. Participants will place their hands on the wall and performed foot stretches with the feet apart, 30 to 50 cm from the wall. Side row, biceps stretch and frontal row. Throwing and receiving, with a distance between 3 to 4 m.
  Interventions: Other: plyometric exercises
- dynamic balance group control group (Other): Control group will be given with the standard physical therapy intervention that includes progressive resistance training that will be performed using weights, two sets of 10 repetitions will be given for each muscle group, resistance will be increased by ½ Kg as children are able to complete without undue stresses); balance exercises (stand on a balance board, one-leg stance, heal-to-toes stance, walking on balance board, walking on a balance beam, walking on a line, and walking on the inclined surface); flexibility exercises
  Interventions: Other: dynamic balance group control group

INTERVENTIONS:
Other: plyometric exercises — Experimental group will be given baseline exercises along with plyometric exercises such as Vertical jump, run and jump, drop jump (jump height between 40 and 50 cm) drop jump and horizontal jump with same height from 3rd week.particepents perform exercises carrying medicine balls. Participants will place their hands on the wall and performed foot stretches with the feet apart, 30 to 50 cm from the wall. Side row, biceps stretch and frontal row. Throwing and receiving, with a distance between 3 to 4 m.
  Other Names: Balance
  Arms: plyometric group
Other: dynamic balance group control group — Control group will be given with the standard physical therapy intervention that includes progressive resistance training that will be performed using weights, two sets of 10 repetitions will be given for each muscle group, resistance will be increased by ½ Kg as children are able to complete without undue stresses); balance exercises (stand on a balance board, one-leg stance, heal-to-toes stance, walking on balance board, walking on a balance beam, walking on a line, and walking on the inclined surface); flexibility exercises
  Arms: dynamic balance group control group

SUMMARY:
Down syndrome is a condition in which a person has an extra chromosome. Typically, a baby is born with 46 chromosomes. Down syndrome is a genetic condition that causes mild to serious physical and developmental problems. Symptoms associated with the syndrome include mental retardation, distinctive facial characteristics, and increased risk for heart defects and digestive problems, which can range from mild to severe.. Early treatment programs can help improve skills. They may include speech, physical, occupational, and/or educational therapy. The aim of the the current study is to determine the effects of plyometric exercise on static and dynamic balance in children with Down syndrome

DETAILED DESCRIPTION:
This will be a randomized controlled trail. After approval from ethical committee, data will be collected from rising sun institute of special education, Lahore. Total sample size will be 20 and there will be two groups. Group A will be given with Standard Physical therapy treatment twice a week for 8 weeks. While group B will be given with plyometric exercises along with standard physical therapy treatment twice a week for 8 weeks. Patients will be evaluated before and after the intervention on Pediatric balance scale, time up and go test, five times sit to stand. Data will be analyzed on SPSS 26.0 and necessary analysis will be done after checking the normality of data.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 12 years of age both genders will be included.
* Children with medical diagnosis of DS.
* Able to follow the command

Exclusion Criteria:

* Recent injury to lower extremities.
* Children with cerebral palsy and other neuromuscular disease will be excluded.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Balance and standing | 8 weeks
  Paediatric berg balance scale

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Khalid, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elnaggar RK. Effects of plyometric exercises on muscle-activation strategies and response-capacity to balance threats in children with hemiplegic cerebral palsy. Physiother Theory Pract. 2022 Sep;38(9):1165-1173. doi: 10.1080/09593985.2020.1833389. Epub 2020 Oct 12. PMID 33044886